CLINICAL TRIAL: NCT06488937
Title: Determinants of Orofacial Pain and Temporomandibular Disorders in People With Rheumatoid Arthritis
Brief Title: Biomarkers Associated With Temporomandibular Disorders in Patients With Rheumatoid Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Collaborators: University of Rijeka Faculty of Dental Medicine (Unknown)
Responsible Party: Principal Investigator, Matea Dozet, DMD, Josip Juraj Strossmayer University of Osijek
Other Study IDs: 01-000-00-678-4./2019.; IP2-FDMZ-2021 (Other Grant/Funding Number: Faculty of dental medicine and health Osijek, Josip Juraj Strossmayer University Osijek)
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Temporomandibular Disorders; Rheumatoid Arthritis
Keywords: RA; rheumatoid arthritis; TMDs; temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood and saliva will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients: Patients that are diagnosed rheumatoid arthritis by their rheumatologist according to the 2010 European League Against Rheumatism/American College of Rheumatology classification criteria.
- Contorol group: The control group will be patients recruited from among regular patients visiting hospital for annual systematic examination in the same hospital.

SUMMARY:
The goal of this observational study is to determinate temeporomandibular disorders (TMDs) and levels of biomarkers in 30 rheumatoid arthritis patients and 30 healthy controls.

Aims are:

* to determine TMDs symptoms in both groups using a validated Reasearch Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) protocol
* to determine levels of interleukin-4 (IL-4), interleukin-18 (IL-18) and interferon-gamma (IFN-γ) in saliva and serum in RA patients and control group
* to determine levels of biomarkers (Ca, Mg, P, AST,ALT,ALP,GGT,urate) in serum of RA patients and control group
* investigate the correlation between cytokines level in saliva and serum
* to determine the effect of TMDs on cytokine and biomarker levels Participants will be clinicaly examined by DMD in accordance with the RDC/TMD guidelines to receive both Axis I and Axis II diagnoses. After examination participants would be asked for saliva and blood sample.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is chronic inflammatory autoimmune disease characterized by symmetrical peripheral polyarthritis with consequent joint destruction. Predominantly affecting wrist and foot joints, RA can also affect temporomandibular joint (TMJ) causing temporomandibular disorders (TMDs). 4-80% of RA patients suffer from TMDs.

It remains unclear why some RA patients do not have TMDs and don't suffer from orofacial pain, depression and somatization. The present study was therefore designed to explore the level of cytokines and biochemical parameters from saliva and serum in RA patients and control participants to examine their correlation with TMDs. Study results could provide valuable insights for the understanding of the orofacial pain and depression onset in RA patients Participants would be examined by a non-blinded examiner with knowledge to which group the patient was in. After intraoral examination Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) will be used as an international diagnostic protocol for TMDs. Assessment included clinical examination of TMJs and masticatory muscles with measurement of mandibular dynamics. The participants will be requested to spit 2 mL of unstimulated saliva into a sterile tube with their head slightly bended forward. Saliva samples were stored at -20℃ until analysis. Blood samples will be collected in Vacutaners. Serum calcium (Ca), magnesium (Mg), phosphate (P), uric acid, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) and gamma-glutamyltransferase (GGT) were measured up to 6 hours after collection. Serum aliquots were stored at -20℃ until cytokine analysis. An Invitrogen assays were used to analyze salivary and serum concentration of IL-4,IL-18 and IFN-γ.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
* Patients diagnosed with RA according to 2010 ACR-EULAR RA criteria.

Exclusion Criteria:

* Refusal to sign informed consent form
* Diagnosed chronic systemic disease
* Any infection including TB, HIV, Hepatitis B or C
* Malignancy
* Pregnancy
* Smokers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with RA were recruited during their routine monitoring by rheumatologists.
  The control group were recruited from among regular patients visiting hospital for annual systematic examination.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
levels of cytokines IL-4, IL-18, IFN-γ in serum | baseline
  Invitrogen assays will be used for multicomplex quantitative analysis of inflammatory mediators. The entire protocol will be carried out according to the instructions of the manufacturer of Thermofischer Scientific
levels of cytokines IL-4, IL-18, IFN-γ in saliva | baseline
  Invitrogen assays will be used for multicomplex quantitative analysis of inflammatory mediators. The entire protocol will be carried out according to the instructions of the manufacturer of Thermofischer Scientific
levels of calcium (Ca), magnesium (Mg), phosphate (P), uric acid, alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) and gamma- glutamyltransferase (GGT) in serum | baseline
  measured up to 6 hours after collection on Roche Cobas c501 biochemistry analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Thalassoterapia Opatija, Specijalna bolnica za medicinsku rehabilitaciju bolesti srca, pluća i reumatizma, Opatija, Rijeka, Croatia

REFERENCES:
- [Result] Mesic VF, Laskarin AM, Kehler T, Spalj S, Dozet M, Pavicic DK. Characteristics of Temporomandibular Disorders and Orofacial Pain in Individuals with Rheumatoid Arthritis. Int J Prosthodont. 2023 Nov 1;36(5):630-636. doi: 10.11607/ijp.8145. PMID 36484668